CLINICAL TRIAL: NCT05656820
Title: Prospective Cohort Study on Imaging Genetics of Bicuspid Aortic Valve
Brief Title: Bicuspid Echocardiac Study Team（BEST）
Acronym: BEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suzhou Municipal Hospital (Other)
Responsible Party: Principal Investigator, Mo Zhou, Attending physician, Suzhou Municipal Hospital
Other Study IDs: GSKY20220407
Record Dates: First submitted 2022-11-28; First posted 2022-12-19 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Bicuspid Aortic Valve Disease
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Chinese Bicuspid Aortic Valve (BAV) Ultrasound imaging cohort study is a Chinese BAV ultrasound imaging cohort study. At present, a retrospective study cohort involving more than 30 hospitals has been established. The prospective multi-center study of BAV is expected to include and follow up 200 outpatients and inpatients with BAV. The clinical, ultrasound imaging and treatment parameters of the patients are collected and the patients are followed up for 2 years. To analyze the prognostic characteristics of BAV patients and establish a Chinese BAV database. The primary endpoint was all-cause death, and the secondary endpoints were heart failure, angina, severe aortic stenosis, severe aortic insufficiency, ascending aortic diameter ≥50mm, and surgery (surgical and interventional). According to the different pathological types of aortic valve in different types of BAV, ultrasound imaging was used to evaluate the different forms of valvular leaflet lesions and prognosis. Finally, it provides a basis for the prognosis, treatment method, treatment timing and treatment plan selection of BAV patients, and lays a foundation for the mechanism study of BAV arterial lesions and the establishment of risk model for the prognosis of BAV patients.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound or other imaging tests to diagnose patients with BAV

Exclusion Criteria:

* Patients with TAV or/and have significant aortic valve calcification
* Those deemed unsuitable for enrollment by clinicians (e.g., end-stage patients, mentally ill patients, non-cooperating patients, etc.)
* Those who do not agree to be included

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient, inpatient, physical examination or community referral patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Diameter of ascending aorta | baseline; once a year; through study completion.
  Diameter of ascending aorta shall be taken using leading edge-to-leading edge convention at end diastole.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Municipal Hospital, Suzhou, China